CLINICAL TRIAL: NCT02303990
Title: RADVAX: A Stratified Phase I Trial of Pembrolizumab With Hypofractionated Radiotherapy in Patients With Advanced and Metastatic Cancers
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Abramson Cancer Center at Penn Medicine (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: UPCC 40914
Record Dates: First submitted 2014-11-26; First posted 2014-12-01 (Estimated); Results first posted 2021-04-22 (Actual); Last update posted 2021-05-12 (Actual); Status verified 2021-04

CONDITIONS: Metastatic Cancers
MeSH Terms: conditions — Neoplasms | interventions — pembrolizumab; Radiotherapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Single arm (Experimental): Hypofractionated RT and Pembro
  Interventions: Drug: Pembrolizumab; Radiation: Radiotherapy

INTERVENTIONS:
Drug: Pembrolizumab
Radiation: Radiotherapy

SUMMARY:
Phase I clinical trial of hypofractionated radiotherapy to an isolated index lesion in combination with the PD-1 inhibitor, Pembrolizumab in patients with metastatic cancers who have failed anti-PD-1 therapy (melanoma and NSCLC) and patients with metastatic cancers who have have progressed after at least one regimen of systemic therapy (breast, pancreas, and other).

ELIGIBILITY:
Inclusion Criteria:

* Be willing and able to provide written informed consent/assent for the trial.
* Be 18 years of age on day of signing informed consent.
* Histologically confirmed diagnosis of cancer as per the cohort specifications
* Stage IV cancer by AJCC staging criteria (except for pancreatic cancer cohort)
* Locally advanced or metastatic pancreatic cancer for the pancreatic cancer cohort
* Progression of disease while on anti-PD-1 or anti-PD-L1 therapy for melanoma and NSCLC patients. For this group, patients must met the following criteria:

  1. Received at least 2 doses of an anti-PD1 or anti-PD-L1 therapy
  2. Had progressive disease documented radiologically by RECIST v1.1 criteria.
* Progression or refractory disease to at least one regimen of therapy for metastatic disease in the breast and pancreatic cancer cohorts
* Presence of an index lesion > 1 cm amenable to hypofractionated radiotherapy
* Patients who have metastatic cancer must have at least one lesion that is outside the radiation field that measures greater than one cm that can be followed by RECIST 1.1. This lesion, if it is close to the radiated lesion, must receive no more than 10% of the dose prescribed to the target lesion.
* Have provided tissue from an archival tissue sample or newly obtained core or excisional biopsy of a tumor lesion.
* Have a performance status of 0 or 1 on the ECOG Performance Scale.
* Ability to tolerate hypofractionated radiation therapy (e.g. lie flat and hold position)
* Demonstrate adequate organ function , all screening labs should be performed within 14 days of treatment initiation.
* Adequate Organ Function Laboratory Values System Laboratory Value Hematological Absolute neutrophil count (ANC) ≥1,500 /mcL Platelets ≥100,000 / mcL Hemoglobin ≥9 g/dL or ≥5.6 mmol/L Renal Serum creatinine OR Measured or calculateda creatinine clearance (GFR can also be used in place of creatinine or CrCl)

  * 1.5 X upper limit of normal (ULN) OR

    ≥60 mL/min for subject with creatinine levels > 1.5 X institutional ULN Hepatic Serum total bilirubin
  * 1.5 X ULN OR Direct bilirubin ≤ ULN for subjects with total bilirubin levels > 1.5 ULN AST (SGOT) and ALT (SGPT)
  * 2.5 X ULN OR
  * 5 X ULN for subjects with liver metastases Creatinine clearance should be calculated per institutional standard
* Female subject of childbearing potential should have a negative urine or serum pregnancy within 72 hours prior to receiving the first dose of study medication. If the urine test is positive or cannot be confirmed as negative, a serum pregnancy test will be required.
* Female subjects of childbearing potential should be willing to use 2 methods of birth control or be surgically sterile, or abstain from heterosexual activity for the course of the study through 120 days after the last dose of study medication. Subjects of childbearing potential are those who have not been surgically sterilized or have not been free from menses for > 1 year.
* Male subjects should agree to use an adequate method of contraception starting with the first dose of study therapy through 120 days after the last dose of study therapy.

Exclusion Criteria

* The subject must be excluded from participating in the trial if the subject:
* Is currently participating in or has participated in a study of an investigational agent or using an investigational device within 4 weeks of the first dose of treatment.
* Has a diagnosis of immunodeficiency or is receiving systemic steroid therapy or any other form of immunosuppressive therapy within 7 days prior to the first dose of trial treatment. Systemic steroids administered specifically as a premedication for chemotherapy infusion or radiotherapy are allowed.
* Has had a prior monoclonal antibody within 4 weeks prior to study Day 1 or who has not recovered (i.e., ≤ Grade 1 or at baseline) from adverse events due to agents administered more than 4 weeks earlier.
* Has had prior chemotherapy, targeted small molecule therapy, or radiation therapy within 2 weeks prior to study Day 1 or who has not recovered (i.e., ≤ Grade 1 or at baseline) from adverse events due to a previously administered agent.
* Note: Subjects with ≤ Grade 2 neuropathy are an exception to this criterion and may qualify for the study.
* Note: If subject received major surgery, they must have recovered adequately from the toxicity and/or complications from the intervention prior to starting therapy.
* A history of prior radiotherapy that precludes delivery of hypofractionated radiotherapy
* Has a known additional malignancy that is progressing or requires active treatment. Exceptions include basal cell carcinoma of the skin, squamous cell carcinoma of the skin, or in situ cervical cancer that has undergone potentially curative therapy.
* Has known active central nervous system (CNS) metastases and/or carcinomatous meningitis. Subjects with previously treated brain metastases may participate provided they are stable (without evidence of progression by imaging for at least four weeks prior to the first dose of trial treatment and any neurologic symptoms have returned to baseline), have no evidence of new or enlarging brain metastases, and are not using steroids for at least 7 days prior to trial treatment.
* Has an active automimmune disease requiring systemic treatment within the past 3 months or a documented history of clinically severe autoimmune disease, or a syndrome that requires systemic steroids or immunosuppressive agents. Subjects with vitiligo or resolved childhood asthma/atopy would be an exception to this rule. Subjects that require intermittent use of bronchodilators or local steroid injections would not be excluded from the study. Subjects with hypothyroidism stable on hormone replacement or Sjogren's syndrome will not be excluded from the study.
* Has evidence of interstitial lung disease or active, non-infectious pneumonitis.
* Has an active infection requiring systemic therapy. Has a history or current evidence of any condition, therapy, or laboratory abnormality that might confound the results of the trial, interfere with the subject's participation for the full duration of the trial, or is not in the best interest of the subject to participate, in the opinion of the treating investigator.
* Has known psychiatric or substance abuse disorders that would interfere with cooperation with the requirements of the trial.
* Is pregnant or breastfeeding, or expecting to conceive or father children within the projected duration of the trial, starting with the pre-screening or screening visit through 120 days after the last dose of trial treatment.
* Has a known history of Human Immunodeficiency Virus (HIV) (HIV 1/2 antibodies).
* Has known active Hepatitis B (e.g., HBsAg reactive) or Hepatitis C (e.g., HCV RNA [qualitative] is detected).
* Has received a live vaccine within 30 days prior to the first dose of trial treatment.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 59 (Actual)
Dates: Start 2015-01-08 (Actual); Primary Completion 2018-12 (Actual); Study Completion 2019-12-31 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Amit Maity, MD, PhD, Principal Investigator — Abramson Cancer Center at Penn Medicine
Locations (1):
- Abramson Cancer Center of the University of Pennsylvania, Philadelphia, Pennsylvania, United States

REFERENCES:
- [Derived] Maity A, Mick R, Huang AC, George SM, Farwell MD, Lukens JN, Berman AT, Mitchell TC, Bauml J, Schuchter LM, O'Hara M, Lin LL, Demichele A, Christodouleas JP, Haas NB, Patsch DM, Hahn SM, Minn AJ, Wherry EJ, Vonderheide RH. A phase I trial of pembrolizumab with hypofractionated radiotherapy in patients with metastatic solid tumours. Br J Cancer. 2018 Nov;119(10):1200-1207. doi: 10.1038/s41416-018-0281-9. Epub 2018 Oct 15. PMID 30318516

RESULTS

PARTICIPANT FLOW:
Groups:
- Single Arm: Hypofractionated RT and Pembro
  Pembrolizumab
  Radiotherapy
Period: Overall Study
Arm/Group | Single Arm
Started | 59
Completed | 59
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Single Arm
Number analyzed (Participants) | 59
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 32
  >=65 years | 27
Age, Continuous [Median (Full Range); unit: years] | 60 [27 to 90]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 35
  Male | 24
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 59
  Not Hispanic or Latino | 0
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 3
  White | 56
  More than one race | 0
  Unknown or Not Reported | 0

OUTCOME MEASURES:

1. Primary Outcome: Number of Adverse Events
Time Frame: 2 years
Measure: Number; unit: Adverse Events
Arm/Group | Single Arm
Number analyzed (Participants) | 59
Adverse Events | 428

ADVERSE EVENTS:
Time Frame: 2 years
Arm/Group | Single Arm
All-Cause Mortality (participants affected / at risk) | 8/59
Serious Adverse Events (participants affected / at risk) | 21/59
Other Adverse Events (participants affected / at risk) | 55/59
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Single Arm (N=59)
Death (General disorders) | 8
Anemia (Blood and lymphatic system disorders) | 1
Not Otherwise Specified (General disorders) | 6
Dehydration (Gastrointestinal disorders) | 1
Dizziness (General disorders) | 1
Fatigue (General disorders) | 1
Fever (General disorders) | 1
Hypotension (Cardiac disorders) | 1
Nausea (General disorders) | 1
Respiratory Failure (Respiratory, thoracic and mediastinal disorders) | 1
Sepsis (General disorders) | 1
Small Intestine Obstruction (Gastrointestinal disorders) | 1
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Single Arm (N=59)
Not otherwise specified (General disorders) | 24
Abdominal distension (General disorders) | 1
Abdominal Pain (General disorders) | 11
Alkaline phosphatase increased (General disorders) | 1
Alopecia (General disorders) | 1
Anemia (General disorders) | 1
Anorexia (General disorders) | 21
Anxiety (General disorders) | 5
Arthralgia (General disorders) | 2
Anrhritis (General disorders) | 1
Ataxia (General disorders) | 1
Back Pain (General disorders) | 5
Bloating (General disorders) | 7
Blurred vision (General disorders) | 2
Bone Pain (General disorders) | 3
Bronchospasm (General disorders) | 1
Bruising (General disorders) | 2
Chest wall pain (General disorders) | 1
Chills (General disorders) | 4
Colitis (General disorders) | 1
Confusion (General disorders) | 5
Conjunctivitis (General disorders) | 1
Constipation (General disorders) | 13
Cough (General disorders) | 15
Dehydration (General disorders) | 5
Depressed Level of Consciousness (General disorders) | 1
Depression (General disorders) | 8
Dermatitis Radiation (General disorders) | 1
Diarrhea (General disorders) | 6
Dizziness (General disorders) | 5
Dry Mouth (General disorders) | 2
Dysgeusia (General disorders) | 2
Dyspepsia (General disorders) | 8
Dysphagia (General disorders) | 3
Dyspnea (General disorders) | 9
Edema limbs (General disorders) | 6
Erythema Multiforme (General disorders) | 1
Esphagitis (General disorders) | 1
Extraocular muscle disorder (General disorders) | 1
Facial muscle weakness (General disorders) | 1
Fall (General disorders) | 3
Fatigue (General disorders) | 28
Fecal Incontinence (General disorders) | 1
Fever (General disorders) | 6
Flank pain (General disorders) | 2
Flatulence (General disorders) | 2
Flu like symptoms (General disorders) | 1
Flushing (General disorders) | 1
Gastritis (General disorders) | 1
Gastroesophageal reflux disease (General disorders) | 3
Generalized muscle weakness (General disorders) | 2
Hand-and-foot syndrome (General disorders) | 1
headache (General disorders) | 6
Hematuria (General disorders) | 1
Hoarseness (General disorders) | 1
Hot flashes (General disorders) | 1
Hypercalcemia (General disorders) | 1
Hypoxia (General disorders) | 1
Ileus (General disorders) | 1
Insomnia (General disorders) | 6
Localized Edema (General disorders) | 3
Lymphocyte count decreased (General disorders) | 2
Muscle weakness upper limb (General disorders) | 1
Myalgia (General disorders) | 1
Nausea (General disorders) | 22
Neck Edema (General disorders) | 1
Neck pain (General disorders) | 3
Non-cardiac chest pain (General disorders) | 2
pain (General disorders) | 3
Pain in extremity (General disorders) | 3
palpitations (General disorders) | 3
paresthesia (General disorders) | 2
Pelvic pain (General disorders) | 1
Peripheral sensory neuropathy (General disorders) | 1
Pleural effusion (General disorders) | 4
portal vein thrombosis (General disorders) | 1
pruritus (General disorders) | 5
scalp pain (General disorders) | 2
sepsis (General disorders) | 1
Sinusititis (General disorders) | 1
Sore throat (General disorders) | 1
Upper respiratory infection (General disorders) | 5
Urinary tract infection (General disorders) | 2
Voice alteration (General disorders) | 1
Vomiting (General disorders) | 8
Weight loss (General disorders) | 3
Wheezing (General disorders) | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2017-08-07): https://cdn.clinicaltrials.gov/large-docs/90/NCT02303990/Prot_SAP_000.pdf